CLINICAL TRIAL: NCT02358577
Title: Early Exercise in Critically Ill Youth and Children, a preLiminary Evaluation.
Brief Title: Early In-bed Cycling in Critically Ill Children
Acronym: wEECycle
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-530
Record Dates: First submitted 2015-01-22; First posted 2015-02-09 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cycle ergometry (Experimental): Participants will receive In-bed cycling for 30 minutes per day in addition to Usual Care, until the physiotherapist deems that the patient is mobilizing well, or a maximum of 7 days (whichever comes first).
  Interventions: Device: In-bed cycling
- Usual care (Active Comparator): Usual care physiotherapy will be applied to patients in the control arm, according to the unit specific guidelines for early mobilization
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: In-bed cycling — In-bed cycling will be applied using a cycle ergometer (RT300 Supine Cycle Ergometer) for 30 minutes per day in addition to Usual Care, until the physiotherapist deems that the patient is mobilizing well, or a maximum of 7 days (whichever comes first). This cycle ergometer is specifically designed for pediatric use, and can be applied to facilitate lower or upper limb cycling. The intervention will be applied by a trained physiotherapist and/or clinician. Pre-defined Safety Criteria for interrupting or aborting the intervention will be observed. Qualitative interviews will be conducted with a health care provider, the patient where possible, and a family caregiver following the intervention period.
  Other Names: Cycle ergometry
  Arms: Cycle ergometry
Other: Usual Care — Usual care physiotherapy will be applied to patients in the control arm, according to the unit specific guidelines for early mobilization. Qualitative interviews will be conducted with a health care provider, the patient where possible, and a family caregiver following the intervention period.
  Arms: Usual care

SUMMARY:
To evaluate the feasibility of conducting a randomized controlled trial (RCT) evaluating the efficacy of early in-bed cycling in addition to usual care physiotherapy, compared to usual care physiotherapy, on functional recovery in critically ill children.

DETAILED DESCRIPTION:
This is a single centre, Pilot RCT that will evaluate in-bed cycling in addition to usual care physiotherapy, compared to usual care physiotherapy, on functional recovery in critically ill children. We will conduct a qualitative substudy to evaluate caregiver impressions of the intervention, and to understand barriers and facilitators to implementing early mobilization in critically ill children.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 3 years to < 18 years;
2. Limited to bed-rest or bed mobility at time of screening
3. expected PICU stay for an additional 48 hours minimum, at time of screening
4. informed consent and or assent where appropriate;
5. agreement of the most responsible PICU physician.

Exclusion Criteria:

1. Contraindications: e.g. Hemodynamic instability, unstable or uncontrolled arrhythmia, ICP, unstable airway, unstable fractures/spine
2. Contraindication to mobilizing upper/lower limbs, e.g. femoral sheath
3. Cycle ergometer does not fit body dimensions
4. Already mobilizing well/expected to mobilize out of bed within 24h
5. not expected to survive current admission - i.e. predicted hospital mortality of > 90%;

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Feasibility - enrolment (75% consent rate target) and protocol adherence | 7 days
  Feasibility is defined as the ability to screen and enrol eligible patients (75% consent rate target).Protocol adherence will be defined as the ability to apply in-bed cycling intervention within 24 hours of consent, and the ability to apply 30 minutes of in-bed cycling daily during week days. We will also measure the rates and reasons for protocol suspensions, violations and study withdrawal.

SECONDARY OUTCOMES:
Adverse event rate | 7 days
  Adverse event rates, physiological parameters prior to, during and after the intervention, discomfort or pain related to the study intervention (as measured by validated pediatric scores).

OTHER OUTCOMES:
Functional outcome (functional recovery, as measured by the Pediatric Overall Performance (POPC), the Pediatric Cerebral Performance Category (PCPC) Scores, and the Pediatric Disability Inventory) | PCCU discharge, 3 and 6 months post PCCU discharge
  We will assess functional recovery at 3 and 6 months (as measured by the Pediatric Overall Performance (POPC), the Pediatric Cerebral Performance Category (PCPC) Scores, and the Pediatric Disability Inventory)
Workload (physiotherapist and nursing workload, as measured by set up and take down times) | 7 days
  We will assess the physiotherapist and nursing workload in both groups
Organ Dysfunction severity as measured by PELOD-2 | 30 days
  organ dysfunction severity progression will be measured by the Pediatric Logistic Organ Dysfunction score (PELOD-2)
PCCU-acquired morbidities | 30 days
  Incidence of PCCU-acquired weakness, pressure ulcers, delirium, sedation withdrawal and delirium
Mortality | 6 months
  PCCU, hospital, 3 and 6 month mortality
Duration of Mechanical Ventilatory support | 30 days
  The number of days on mechanical ventilatory support, and the number of days alive and free of mechanical ventilatory support at 30 days
Length of stay | 30 days
  The length of Paediatric intensive care unit and hospital stay, will be measured
Caregiver perception | 7 days
  Caregiver impressions of early mobilization interventions, and barriers and facilitators to early mobilization in critically ill children

CONTACTS AND LOCATIONS:
Overall Officials: Karen Choong, MB, BCh, MSc, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada